CLINICAL TRIAL: NCT05673967
Title: A Study to Characterize Treatment Patterns and Real-World Outcomes in Heavily Pretreated Patients With Relapsed and Refractory Multiple Myeloma (RRMM) and Similar Clinical Characteristics to Patients in the Phase 2 Cohort 2 of the R5458-ONC-1826 Trial
Brief Title: Real-World Clinical Outcomes in Patients With Relapsed/Refractory Multiple Myeloma
Status: Completed | Type: Observational
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: R5458-ONC-21101
Record Dates: First submitted 2022-12-21; First posted 2023-01-06 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Relapsed and Refractory Multiple Myeloma (RRMM)
Keywords: Real-World Outcomes; Multiple Myeloma (MM); Objective response rate (ORR); Triple-class exposed (TCE); Triple-class refractory (TCR); Progression-free survival (PFS); Overall survival (OS)
MeSH Terms: conditions — Recurrence; Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: Real-world (RW) patients with RRMM who have either at least three prior lines of therapy (LOT) and are triple-class exposed (3L+/TCE), or are triple-class refractory (TCR), meet similar inclusion/exclusion criteria used to establish phase 2 cohort 2 of the R5458-ONC-1826 trial, and are initiating currently available therapies.
  Interventions: Other: Non-Interventional

INTERVENTIONS:
Other: Non-Interventional — No study treatment will be administered on this study.

SUMMARY:
Primary Objective:

1. To describe the distribution of treatment regimens and objective response rate (ORR) in a Benchmark Cohort of real-world patients with relapsed/refractory multiple myeloma (RRMM) who initiate treatment after meeting the following criteria: (1) have either (a) at least three prior lines (3L) and are triple-class exposed (TCE), or (b) are triple-class refractory (TCR), and (2) meet similar inclusion/exclusion criteria to patients in phase 2 cohort 2 of the R5458-ONC-1826 (NCT03761108) trial.

Secondary Objectives:

1. To describe additional outcomes (duration of response [DOR], progression-free survival [PFS], overall survival [OS], and time to next treatment [TTNT]) in the same Benchmark Cohort population described in the primary objective.
2. To describe distribution of treatment regimens, ORR, DOR, PFS, OS, and to compare ORR, PFS, OS, and TTNT in an Analysis Cohort consisting of real-world patients derived from the Benchmark Cohort described above who are weighted to align with the characteristics of patients in phase 2 cohort 2 of the R5458-ONC-1826 (NCT03761108) trial. Comparative analyses of PFS and OS will be performed conditional on sufficient maturity of survival data in the R5458-ONC-1826 (NCT03761108) trial at the time of analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Eastern Cooperative Oncology Group (ECOG) performance status ≤1 at baseline
2. Confirmed diagnosis of active MM by IMWG diagnostic criteria
3. Have myeloma that is response-evaluable with measurable disease by M-protein in serum or urine as specified in the IMWG response criteria.
4. Triple-class exposed or refractory

Exclusion Criteria:

1. Diagnosis of plasma cell leukemia, primary systemic light-chain amyloidosis (excluding myeloma-associated amyloidosis), Waldenström macroglobulinemia, or polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin (POEMS) changes syndrome
2. Known MM brain lesions or meningeal involvement
3. History of neurodegenerative condition, central nervous system (CNS) movement disorder, or seizure
4. Cardiac ejection fraction <40% by echocardiogram or multi-gated acquisition scan (MUGA) (or a diagnosis of congestive heart failure, cardiomyopathy, or valvular heart disease as a potential proxy)
5. Continuous systemic corticosteroid treatment with more than 10 mg per day of prednisone or anti-inflammatory equivalent
6. Live or live attenuated vaccines
7. Treated with B-cell maturation antigen (BCMA)-directed immunotherapies (BCMA antibody-drug conjugates are not excluded).

Note: Other protocol-defined Inclusion/Exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with RRMM who have either at least three prior lines of therapy (LOT) and are triple-class exposed (3L+/TCE), or are triple-class refractory (TCR).
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2024-09-12 (Actual); Study Completion 2025-03-28 (Actual)

PRIMARY OUTCOMES:
Proportion of patients exposed to each type of regimen by line of therapy (LOT) | Up to 6 years
  Distribution of treatment regimens
Proportion of patients with objective response rate (ORR) | Up to 6 years
  Defined as stringent complete response (sCR), complete response (CR), very good partial response (VGPR), or partial response (PR)

SECONDARY OUTCOMES:
Duration of response (DOR) | Up to 6 years
  Defined as time from the date of the first documented response (best overall response of sCR, CR, VGPR, PR) until the first date of progressive disease (PD) by International Myeloma Working Group (IMWG) or death due to any cause, whichever occurs first.
Progression-free survival (PFS) | Up to 6 years
  Defined as time from the start of study treatment until the first date of PD by IMWG, or death due to any cause, whichever occurs first.
Overall survival (OS) | Up to 6 years
  OS is measured from the start of study treatment until death due to any cause.
Time to next treatment (TTNT) | Up to 6 years
  Defined as time from the start of study treatment until the initiation of the subsequent LOT.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (1):
- Regeneron Research Facility, Tarrytown, New York, United States